CLINICAL TRIAL: NCT03397563
Title: Continuous Positive Airway Pressure as a Potential New Treatment for Cluster Headache - a Randomized Controlled Crossover Study
Brief Title: Continuous Positive Airway Pressure as a Potential New Treatment for Cluster Headache
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017/1491
Record Dates: First submitted 2018-01-04; First posted 2018-01-12 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Cluster Headache; Chronic Disease
Keywords: Continuous Positive Airway Pressure; Sleep Apnea, Obstructive; Polysomnography
MeSH Terms: conditions — Cluster Headache; Chronic Disease; Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP treatment (Experimental): Continuous Positive Airway Pressure (CPAP)
  Interventions: Device: Continuous Positive Airway Pressure; Device: sham Continuous Positive Airway Pressure
- Sham-CPAP treatment (Sham Comparator): sham Continuous Positive Airway Pressure (sham-CPAP)
  Interventions: Device: Continuous Positive Airway Pressure; Device: sham Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — standard automatic CPAP machine set on optimal automatic pressure
  Other Names: CPAP
Device: sham Continuous Positive Airway Pressure — CPAP machine with pressure set below effective impact, i.e. low pressure of 4 cm H2O and adjustment of the ventilation mask
  Other Names: sham-CPAP

SUMMARY:
Cluster headache is also called suicide headache due to excruciating nocturnal attacks. There are few treatment options available. Inhalation of oxygen has shown to abort the attacks.

Continuous positive airway pressure (CPAP) is a machine used during sleep to treat respiratory failure. Automatic CPAP machines adjust the air pressure through the night to keep the upper airways patent.

Single reports have shown a high prevalence of obstructive sleep apnea in people suffering from cluster headache, and positive effects of CPAP treatment, but no randomized controlled trial has been conducted so far.

If proven effective CPAP would make an affordable treatment option for many patients within the existing healthcare system.

DETAILED DESCRIPTION:
This is a single center study carried out in collaboration between the neurological, neurophysiological and thoracic departments at St. Olavs Hospital in Trondheim.

Participants will keep sleep and headache diaries in a baseline period of 4 weeks, then receive treatment (CPAP or sham-CPAP at nighttime) during 8 weeks, have a 4 week wash out period followed by a second treatment period of 8 weeks (CPAP or sham-CPAP). Finally there will be follow-up during 1 month.

Throughout the whole study (7 months) participants keep a headache diary. Participants must maintain current preventive and sleep medication regimens during the whole study period, and may use acute medication of choice (sumatriptan, oxygen or other).

Sleep registration in all participants will be done by polysomnography(PSG). An Ultra Wide Band radar/movement sensor device will be used to detect sleep patterns, together with wrist pulse oximetry and wrist actigraphy during PSG and the last week of each treatment period.

Neurophysiologic tests such as temperature and pressure thresholds will be measured before PSG and after each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Fulfils the diagnostic criteria for chronic cluster headache according to ICHD-3 beta 3.1.2.
* is able to separate cluster headache attacks from other types of headache.
* agrees to maintain current preventive headache and sleep medication regimens (no change in type, frequency, or dose) during the whole study period.
* Signed informed consent.

Exclusion Criteria:

* disorders with contraindications for use of continuous positive airway pressure (e.g. unable to remove the ventilation mask due to a movement disorders).
* Nightly cluster headache attacks
* Pregnancy or planned pregnancy
* having had a change in type, dosage or dose frequency of preventive headache or sleep medications < 1 months prior to inclusion.
* Severe depression or other psychiatric disorder that may interfere with the treatment.
* Abuse of alcohol or illicit drugs.
* Other severe chronic pain conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
change from baseline in number of cluster headache attacks per week at week 9-12 | 12 weeks
change from baseline in number of cluster headache attacks per week at week 21-24 | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in the number of nightly cluster attacks per week at week 9-12 | 12 weeks
Change from baseline in the number of nightly cluster attacks per week at week 21-24 | 24 weeks
Change from baseline in cluster headache start time per week at week 9-12 | 12 weeks
Change from baseline in cluster headache start time per week at week 21-24 | 24 weeks
Change from baseline in the number of days with cluster headache per week at week 9-12 | 12 weeks
Change from baseline in the number of days with cluster headache per week at week 21-24 | 24 weeks
Change from baseline in the number of hours with cluster headache per week at week 9-12 | 12 weeks
Change from baseline in the number of hours with cluster headache per week at week 21-24 | 24 weeks
Change from baseline in use of acute treatment per week at week 9-12 | 12 weeks
Change from baseline in use of acute treatment per week at week 21-24 | 24 weeks
Change from baseline in subjective sleep quality in week 12 | 12 weeks
  according to sleep diary
Change from baseline in subjective sleep quality in week 24 | 24 weeks
  according to sleep diary
Change from the night of PSG registration in apnea-hypopnea index (AHI) during sleep to week 12 | 12 weeks
Change from the night of PSG registration in apnea-hypopnea index (AHI) during sleep to week 24 | 24 weeks
Change from the night of PSG registration in oxygen desaturation index (ODI) during sleep to week 12 | 12 weeks
Change from the night of PSG registration in oxygen desaturation index (ODI) during sleep to week 24 | 24 weeks
Change from baseline in heat/cold pain thresholds at week 12 according to thermal test | 12 weeks
Change from baseline in pressure pain thresholds at week 12 according to algometry test | 12 weeks
Change from baseline in heat/cold pain thresholds at week 24 according to thermal test. | 24 weeks
Change from baseline in pressure pain thresholds at week 24 according to algometry test | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geirmund Unsgård, MD PhD prof, Study Director — St. Olavs Hospital; Erling Tronvik, MD PhD, Principal Investigator — Norwegian University of Science and Technology; Lars Jacob Stovner, MD prof, Study Chair — Norwegian Advisory Unit on Headaches
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gravdahl GB, Aakeroy L, Stovner LJ, Engstrom M, Muller KI, Bjork MH, Tronvik E. Continuous positive airway pressure in cluster headache: A randomized, placebo-controlled, triple-blind, crossover study. Cephalalgia. 2023 Jan;43(1):3331024221128273. doi: 10.1177/03331024221128273. PMID 36620891